CLINICAL TRIAL: NCT00741325
Title: Long-term Observational Follow-up Study of a Multicenter, Randomized, Double-blind, Placebo-controlled, Comparative Trial of AMD3100 (240µg/kg) Plus G-CSF (10µg/kg) Versus G-CSF (10µg/kg) Plus Placebo to Mobilize and Collect ≥ 5X 10^6 CD34+ Cells/kg in Non-Hodgkin's Lymphoma Patients for Autologous Transplantation
Brief Title: Long-Term Follow-up Study for Non-Hodgkin's Lymphoma Patients Who Received Study Treatment (Plerixafor or Placebo) in the AMD3100-3101 Study (NCT00103610).
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AMD31003101LTF
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Non-Hodgkin's Lymphoma; Autologous Transplantation
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- G-CSF plus plerixafor: Participants in Study AMD3100-3101 (NCT00103610)underwent mobilization with granulocyte colony-stimulating factor (G-CSF)and received plerixafor, prior to undergoing apheresis.
  Interventions: Drug: granulocyte colony-stimulating factor (G-CSF); Drug: plerixafor
- G-CSF plus placebo: Participants in Study AMD3100-3101 (NCT00103610)underwent mobilization with granulocyte colony-stimulating factor (G-CSF)and received placebo, prior to undergoing apheresis.
  Interventions: Drug: granulocyte colony-stimulating factor (G-CSF); Drug: Placebo

INTERVENTIONS:
Drug: granulocyte colony-stimulating factor (G-CSF)
Drug: plerixafor
  Other Names: Mozobil; AMD3100
  Groups: G-CSF plus plerixafor
Drug: Placebo
  Groups: G-CSF plus placebo

SUMMARY:
This is a long-term observational study of patients that were treated with at least 1 dose of study treatment (plerixafor or placebo) in the AMD3100-3101 protocol (NCT00103610).

DETAILED DESCRIPTION:
This is a long-term observational study of patients who received at least one dose of study treatment (plerixafor or placebo) in a multicenter, randomized, double blind, placebo-controlled investigational study to evaluate granulocyte colony stimulating factor (G-CSF) plus AMD3100 versus G-CSF plus placebo to mobilize and transplant Non-Hodgkin's Lymphoma (NHL) patients (protocol AMD3100-3101 [NCT00103610]). The objective of this study is to assess progression-free survival and overall survival of patients treated with at least 1 dose of study treatment (placebo or plerixafor) for a period of 5 years following the first dose of study treatment (placebo or plerixafor) in protocol AMD3100-3101 (NCT00103610).

ELIGIBILITY:
Inclusion Criteria:

* All patients who received a dose of study treatment (plerixafor or placebo)in protocol AMD3100-3101 (NCT00103610)

Exclusion Criteria:

* No Exclusion Criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the AMD3100-3101 study (NCT00103610) who received at least one dose of study treatment (plerixafor or placebo)
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2006-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival and overall survival of patients treated with at least 1 dose of study treatment (placebo or plerixafor) in protocol AMD3100-3101 (NCT00103610). | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company

REFERENCES:
- [Derived] Micallef IN, Stiff PJ, Nademanee AP, Maziarz RT, Horwitz ME, Stadtmauer EA, Kaufman JL, McCarty JM, Vargo R, Cheverton PD, Struijs M, Bolwell B, DiPersio JF. Plerixafor Plus Granulocyte Colony-Stimulating Factor for Patients with Non-Hodgkin Lymphoma and Multiple Myeloma: Long-Term Follow-Up Report. Biol Blood Marrow Transplant. 2018 Jun;24(6):1187-1195. doi: 10.1016/j.bbmt.2018.01.039. Epub 2018 Feb 2. PMID 29410180